CLINICAL TRIAL: NCT05456802
Title: The Influence of a Symptomatic Coronary Artery and Peripheral Arterial Disease on the Oral-enteral Microbiome and Downstream Microbiome-dependent Metabolites
Brief Title: Effect of Acute Cardiovascular Disease on Microbiome
Acronym: MIAMI
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Chistos Rammos, Professor Dr. med., University Hospital, Essen
Other Study IDs: MIAMI Trial
Record Dates: First submitted 2022-06-30; First posted 2022-07-13 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Microbial Colonization; Coronary Artery Disease; Myocardial Infarction; Acute Coronary Syndrome; Peripheral Arterial Disease; Critical Limb Ischemia
MeSH Terms: conditions — Communicable Diseases; Coronary Artery Disease; Myocardial Infarction; Acute Coronary Syndrome; Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — stool and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Acute Coronary Syndrome (ACS): Patients presenting to the clinic with acute coronary syndrome. This includes: ST-elevation myocardial infarction (STEMI), non-ST-elevation myocardial infarction (NSTEMI) and unstable angina pectoris (UAP) with confirmed diagnosis of coronary artery disease.
  Interventions: Other: Standard of care treatment
- Chronic Coronary Syndrome (CCS): Patients presenting to the clinic with chronic coronary syndrome and confirmed diagnosis of coronary artery disease.
  Interventions: Other: Standard of care treatment
- Critical limb ischemia (CLI): Patients presenting to the clinic with critical limb ischemia. This includes: Resting limb pain (Fontaine III), ulcerations (Fontaine IV) and Ankle brachial index (ABI) < 0,6 and confirmed diagnosis of peripheral artery disease.
  Interventions: Other: Standard of care treatment

INTERVENTIONS:
Other: Standard of care treatment — Standard of care treatment including percutaneous interventions was performed in all participants.

SUMMARY:
Atherosclerotic diseases such as coronary artery disease (CAD) and peripheral arterial disease (PAD) are the leading cause of morbidity and mortality in the industrialized world.

An interaction between the development of atherosclerotic diseases and the oral and enteral microbiome composition has already been demonstrated in the past. The microbiome is a double-edged sword which can convey protective and detrimental cardiovascular effects. While it can promote the development of atherosclerosis through the production of atherogenic metabolites such as trimethylamine N-oxide (TMAO) it can also generate a protective effect through the production of metabolites such as short chain fatty acids (SCFA). Preliminary data suggest that atherosclerotic disease itself can induce a dysbiosis of the microbiome.

Aim of this study is to determine the differences in coronary artery disease and peripheral arterial disease on the oral-enteral microbiome axis and downstream microbiome-dependent metabolites.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* patient consent
* CCS, ACS or CLI
* angiographical confirmed peripheral or coronary artery disease

Exclusion Criteria:

* pregnancy/lactation period
* current antibiotic treatment or in the past 3 months
* chronic inflammatory bowel disease
* short bowel syndrome
* artificial bowel outlet
* persistent diarrhea or vomiting in the past 3 months
* simultaneous participation in another interfering nutrition study
* active chemo or radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years presenting to the clinic with acute coronary syndrome (ACS), chronic coronary syndrome (CCS) or critical limb threatening ischemia (CLI) who can be included into the study within a 24 hours time frame after presentation.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Change of enteral microbiome composition after presentation with ACS/CCS/CLI | Sampling will be performed within 24 hours of presentation to the clinic, at day 3, day 7, day 14 and at day 28 (+/- 2 days) after initial presentation.
  Stool samples are collected at the below mentioned time points. DNA isolation will be performed with consecutive 16S-RNA analysis and cluster analysis.
Change of oral microbiome composition after presentation with ACS/CCS/CLI | Sampling will be performed within 24 hours of presentation to the clinic, at day 3, day 7, day 14 and at day 28 (+/- 2 days) after initial presentation.
  Oral samples are collected at the below mentioned time points. DNA isolation will be performed with consecutive 16S-RNA analysis and cluster analysis.

SECONDARY OUTCOMES:
Change of TMAO serum levels after presentation with ACS/CCS/CLI | Sampling will be performed within 24 hours of presentation to the clinic and at day 28 (+/- 2 days) after initial presentation.
  Blood samples are collected at the below mentioned time points. TMAO serum levels will be measured by ultra-high-performance liquid chromatography-tandem mass spectrometry (UHPLC-MS/MS).
Change of SCFA serum levels after presentation with ACS/CCS/CLI | Sampling will be performed within 24 hours of presentation to the clinic and at day 28 (+/- 2 days) after initial presentation.
  Blood samples are collected at the below mentioned time points. SCFA serum levels will be measured by high-performance liquid chromatography (HPLC).

OTHER OUTCOMES:
Change of left ventricular global longitudinal strain (GLS) after presentation with ACS/CCS/CLI | Echocardiography will be performed within 24 hours of presentation to the clinic and at day 28 (+/- 2 days) after initial presentation.
  Echocardiographical strain analysis will be performed at the below mentioned time points.
Change of inflammatory profile (CRP, PCT, Interleukin panel) after presentation with ACS/CCS/CLI | Sampling will be performed within 24 hours of presentation to the clinic and at day 28 (+/- 2 days) after initial presentation.
  Blood samples are collected at the below mentioned time points.
Change of blood pressure after presentation with ACS/CCS/CLI | Blood pressure measurements will be performed within 24 hours of presentation to the clinic and at day 28 (+/- 2 days) after initial presentation.
  Blood pressure will be measured at the below mentioned time points.
Change of pulse wave velocity (PWV) after presentation with ACS/CCS/CLI | PWV measurements will be performed within 24 hours of presentation to the clinic and at day 28 (+/- 2 days) after initial presentation.
  PWV will be measured at the below mentioned time points.
Change in nitrite metabolism after presentation of ACS/CCS/CLI | Nitrite metabolism will be performed within 24 hours of presentation to the clinic and at day 28 (+/- 2 days) after initial presentation.
  Nitrite metabolism will be assed by chemiluminescence detection (CLD).

CONTACTS AND LOCATIONS:
Overall Officials: Christos Rammos, Prof. Dr., Principal Investigator — University Clinic Essen
Locations (1):
- University of Essen, Clinic of Cardiology and Angiology, Essen, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Messiha D, Lange E, Tratnik A, M Westendorf A, Rinke M, Lenz S, Hendgen-Cotta UB, Buer J, Rassaf T, Rammos C. The influence of acute and chronic coronary syndrome on the gut microbiome and downstream microbiome-derived metabolites-Microbiome in acute myocardial infarction-MIAMI-Trial. Basic Res Cardiol. 2025 Oct;120(5):913-924. doi: 10.1007/s00395-025-01134-9. Epub 2025 Aug 13. PMID 40804540